CLINICAL TRIAL: NCT00344942
Title: A Randomised, Double-blind, French Multi-centre Study, to Evaluate the Efficacy and Tolerance, in Comparison With Placebo, of Nasacort in Chronic Non Allergic and Non Infectious Rhinitis in Adults
Brief Title: Efficacy and Safety Study of Nasacort in Chronic Non Allergic and Non Infectious Rhinitis in Adults
Acronym: RhiCNANI
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: patient's recruitment too difficult
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TRICA_L_00872; EudraCT #: 2006-000059-16
Record Dates: First submitted 2006-06-26; First posted 2006-06-27 (Estimated); Last update posted 2009-12-07 (Estimated); Status verified 2009-12

CONDITIONS: Rhinitis
MeSH Terms: conditions — Rhinitis | interventions — Triamcinolone Acetonide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: triamcinolone acetonide
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: triamcinolone acetonide — 220µg/day or a double spray into each nostril once daily for 12 weeks'treatment
  Arms: 1
Drug: placebo — a double spray into each nostril once daily
  Arms: 2

SUMMARY:
To demonstrate the superiority of the clinical efficacy of 12 weeks' treatment with Nasacort versus placebo in adult patients presenting with Chronic Non Allergic and Non Infectious Rhinitis

ELIGIBILITY:
Inclusion Criteria:

* patient presenting with Chronic Non Allergic and Non Infectious Rhinitis capable of benefiting from corticosteroid therapy administered via the nasal route.
* patient with chronic rhinitis of minimum duration 12 weeks, whether or not consecutive, per year.
* patient with Non Allergic Rhinitis confirmed by negative phadiatop test.
* patient presenting a mean global score for the 5 symptoms >= 5 (nasal obstruction, rhinorrhea, disturbance of sense of smell, sneezing, facial heaviness), or mean score for the 3 main symptoms (nasal obstruction, rhinorrhea, disturbance of sense of smell) >= 5 (mean for 7 days prior to visit V0).
* patient presenting an inflammation score at anterior rhinoscopy or nasal endoscopy >= 4.

Exclusion Criteria:

* patient presenting a nasal polyp
* patient presenting a severe septal deviation which would interfere with insertion of the nasal spray
* patient presenting a nasal cavity tumor
* patient presenting a sinus infection
* patient presenting a history of endonasal surgery
* patient presenting a chronic rhinitis of extrinsic origin (drug-related or food-related rhinitis) or intrinsic origin (hormonal rhinitis, positional rhinitis,atrophic rhinitis, ...)
* patient on a program of intensive sports training
* patient presenting with : cystic fibrosis, pulmonary mycosis, necrotising vascularitis, immotile cilia syndrome, ....
* patient presenting with known immunosuppression, lymphoma
* patient presenting with a known cardiovascular, neurological or other medically significant illness
* patient presenting with known renal failure, with known glaucoma, with known drug addiction
* current antibiotic therapy
* corticosteroids administered in the two months prior to admission
* patient presenting problems of haemostasis (epistaxis), ophthalmic and/or oro-bucco-nasal herpetic infection.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2006-04; Primary Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Mean global score obtained on the basis of 5 evaluations : nasal obstruction, rhinorrhea, disturbed sense of smell, sneezing, facial heaviness. | 7 days prior to each visit

SECONDARY OUTCOMES:
list of undesirable events | during the treatment period

CONTACTS AND LOCATIONS:
Overall Officials: M SEBILLE, Dr, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis, Paris, France